CLINICAL TRIAL: NCT05672212
Title: Effect of Goal-directed Analgesia Using ANI (Analgesia/Nociception Index) During General Anesthesia in Children Undergoing EDAS (Encephaloduroarteriosynangiosis) Surgery for Moyamoya Disease: a Randomized Controlled Trial
Brief Title: Goal-directed Analgesia Using ANI During General Anesthesia in Children With Moyamoya Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2211-149-1381
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Analgesia; Sufentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANI (Analgesia/Nociception Index) monitoring (Experimental)
  Interventions: Device: ANI (Analgesia/Nociception Index) monitoring; Drug: Sufentanil
- Standard monitoring (Active Comparator)
  Interventions: Device: standard monitoring; Drug: Sufentanil

INTERVENTIONS:
Device: ANI (Analgesia/Nociception Index) monitoring — Intraoperative analgesia was provided by injection of sufentanil, which was performed according to ANI monitor.
  Arms: ANI (Analgesia/Nociception Index) monitoring
Device: standard monitoring — Intraoperative analgesia was provided by injection of sufentanil, which was performed according to the clinician's assessment.
  Arms: Standard monitoring
Drug: Sufentanil — Sufentanil

SUMMARY:
Analgesia Nociception Index (ANI) has been proposed for the evaluation of the nociception-antinociception balance in the perioperative period. In pediatric patients with Moyamoay disease, where the management of analgesia may be rendered difficult by pharmacological changes, we hypothesised that the monitoring of analgesia with ANI would reduce intraoperative opioid consumption during EDAS surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients receiving EDAS surgery for Moyamoya disease

Exclusion Criteria:

* ASA (American society of anesthsiologists classification) 4-5
* Emergency surgery
* patients with chronic pain on medication

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-01-04 (Estimated); Study Completion 2025-01-04 (Estimated)

PRIMARY OUTCOMES:
the mean hourly intraoperative sufentanil requirement | from induction of anesthesia to end of operation, about 5 hours

SECONDARY OUTCOMES:
the amount of non-opioids analgesic requirements | from induction of anesthesia to end of operation, about 5 hours
the amount of vasoactive agents requirements | from induction of anesthesia to end of operation, about 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park JB, Kang P, Ji SH, Jang YE, Lee JH, Kim JT, Kim HS, Kim EH. Effects of goal-directed analgesia using the analgesia nociception index in children undergoing surgery for moyamoya disease: A randomised controlled trial. Eur J Anaesthesiol. 2024 Sep 1;41(9):649-656. doi: 10.1097/EJA.0000000000002013. Epub 2024 Jun 3. PMID 38832435